CLINICAL TRIAL: NCT04122469
Title: The Role of Stereo-tActic BoDy RadIotherApy iN Oligo-Progressive MalignanT Disease
Acronym: RADIANT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-6047
Record Dates: First submitted 2019-10-04; First posted 2019-10-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Malignancy; Breast Cancer Metastatic; Genito-urinary
Keywords: SBRT
MeSH Terms: conditions — Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oligo-Progression; GU (Experimental): Receiving SBRT.
  Interventions: Radiation: Stereotactic Body Radiotherapy
- Oligo-metastatic Breast Cancer (Experimental): Receiving SBRT.
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — The purpose of this study is to evaluate the safety, and efficacy of SBRT in this patient population

SUMMARY:
Systemic therapy is the main treatment for patients with metastatic cancers. Oligo-progression has become a recognized entity for metastatic cancer and it is thought that a subset of cancer cells may develop heterogeneity and resistant clones while receiving systemic therapy. This results in overall tumor response but progression in metastatic sites. Current standard is to change systemic therapies. With advancing technologies, stereotactic body radiation therapy is being used to deliver high doses of focused radiation to the disease site, while minimizing risk of injury to the surrounding organs. SBRT is increasingly being used in patients presenting oligo-metastatic disease, and is recognized as having a potential for cure. This study will investigate the use of SBRT for breast and genito-urinary cancer patients with oligo-progression. Patients will be seen before and at the end of treatment and will be followed at 4 month intervals for up to 2 years.

During the visits participants will complete quality of life questionnaires and will have standard of care imaging.

Patients will also have the option to provide blood at baseline, during treatment, and at various follow up time points for analysis of ctDNA

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years accrued at the Princess Margaret Cancer Centre
* 5 or less sites of intra or extra-cranial oligo-progressive, de novo oligo-metastatic, induced oligo-metastatic and repeat oligo-metastatic breast disease amenable to ablative treatment (including but not limited to radiotherapy, surgery, radio-frequency ablation);

  o at least one lesion should be planned for SBRT
* OR 5 or less sites of intra or extra-cranial oligo-progressive prostate, bladder and renal cell carcinomas
* Tumor mass amenable to SABR (≤6cm in size)
* Confirmation of diagnosis:

  * Known/documented prior histological (for all excluding HCC) or radiological diagnosis (for HCC) of:
  * Pathologically confirmed breast cancer OR,
  * Pathologically confirmed GU cancer (such as prostate cancer, bladder cancer, or radiologically or pathologically confirmed RCC).
* For prostate patients only: Known metastatic disease treated with ADT (patients who received other ST as first line treatment of mCSPC would be eligible; eg Docetaxel, Abiraterone…)
* For prostate patients only: Known metastatic CRPC progressing on ST (Docetaxel, Abiraterone, Enzalutamide…)
* For oligo-progressive disease: receiving any form of ST for at least 3 months with (ST breaks are permitted):

  1. Radiographic evidence of ≤3 intra or extra-cranial lesions progressing (including nodal or distant). At least one lesion is suitable for SBRT. Each progressing lesion should fulfill at least 1 of the 3 following criteria for oligo-progression:

     1. Progression of a metastasis according to RECIST 1.1 criteria7
     2. Unambiguous development of a new lesion from the time of scan taken prior to starting ST
     3. Progressive enlargement of a known metastasis on 2 consecutive imaging (CT or MRI) 2-3 months apart, while on ST, with a minimum 5 mm increase in size from baseline.
  2. Remainder of metastatic disease stable or regressing, as per RECIST v1.1, evidenced by >2 consecutive images within the past 4-6 months.
* Able to provide written consent
* ECOG performance status 0-3

Exclusion Criteria:

* ≥6 progressive metastases
* Evidence of spinal cord compression or acute event requiring urgent/emergency radiotherapy
* Prior radiotherapy, with fields overlapping, resulting in excessive doses to organs at risk
* Previous radical RT in the area of OP
* Inability to safely treat all sites of progressing metastases
* Patient cannot tolerate physical set-up required for SBRT
* Treatment plan respecting normal tissue tolerances using dose fractionation specified within the protocol cannot be achieved
* Active bowel obstruction, if treating abdominal/pelvic site
* Neuroendocrine, lymphoma, myeloma or germ cell malignancies
* Familial syndromes: Von Hippel-Lindau disease, Polycystic Kidney Disease, Hereditary Papillary RCC or Tuberous Sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-09-11 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Safety of SBRT in OP malignancies | 24 month period
  To determine the safety of SBRT in OP malignancies over a 24-month follow-up period using CTCAE v5.0.
Efficacy of SBRT in OP malignancies | 24 month period
  To determine the efficacy of SBRT in OP malignancies over a 24-month follow-up period by evaluating progression-free survival. Radiographic local control of irradiated areas and local disease will also be used to determine efficacy by using Response Evaluation Criteria in Solid Tumors (RECIST).
Feasibility of SBRT in OP malignancies | 24 month period
  To determine the feasibility of SBRT in OP malignancies over a 24-month follow-up period using the a quality of life questionnaire (the EORTC QLQ-C30 questionnaire).

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada